CLINICAL TRIAL: NCT05652582
Title: Seroprevalence of SARS-CoV 2 in the Staff of the University Hospitals of Strasbourg
Brief Title: Seroprevalence of Covid-19 in the Staff of the University Hospitals of Strasbourg
Acronym: SeroPrevHUS
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8253
Record Dates: First submitted 2022-12-13; First posted 2022-12-15 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: COVID-19
Keywords: COVID-19; SARS-COV-2; Prevalence of SARS-CoV-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Grand Est region is one of the most affected regions in France during the first wave of the COVID-19 epidemic. A significant increase in the number of patients hospitalized for SARS-CoV 2 infection at the University Hospitals of Strasbourg (HUS) led to a sudden saturation of their capacities. Hospital workers appear to be a population at particular risk for this new infectious agent. The percentage of hospital workers who have been in contact with the virus or have contracted COVID-19 is unknown.

The objective of this work is to determine the prevalence of SARS-CoV-2 positive serologies among hospital staff screened from June 22, 2020 to November 1, 2020 following a screening campaign offering serological testing to all volunteer HUS professionals.

ELIGIBILITY:
Inclusion criteria:

* Adult subject (≥ 18 years of age)
* Hospital staff practicing at HUS who performed SARS-CoV 2 serology in the period from 06/22/2020 to 11/1/2020

Exclusion criteria:

- Subject not meeting inclusion criteria

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Hospital staff practicing at HUS who performed SARS-CoV 2 serology in the period from 06/22/2020 to 11/1/2020
Sampling Method: Non-Probability Sample
Enrollment: 5694 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2022-04-24 (Actual); Study Completion 2022-06-24 (Actual)

PRIMARY OUTCOMES:
To determine the positive seroprevalence of SARS-CoV-2 among hospital staff screened from June 22, 2020 to November 1, 2020 | Files analysed retrospectively from June 22, 2020 to November 1, 2020 will be examined
  Seroprevalence will be estimated by calculating the rate of seropositive subjects with its 95% confidence interval

CONTACTS AND LOCATIONS:
Locations (1):
- Service Laboratoire de Virologie - PTM - CHU de Strasbourg - France, Strasbourg, France